CLINICAL TRIAL: NCT01655251
Title: Video Discharge Instructions for Fever and ED Recidivism
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Connecticut Children's Medical Center (Other)
Responsible Party: Principal Investigator, Sharon Smith, ED Research Director, Connecticut Children's Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 10-098-CCMC
Record Dates: First submitted 2012-07-30; First posted 2012-08-01 (Estimated); Results first posted 2025-10-14 (Actual); Last update posted 2025-10-14 (Actual); Status verified 2025-09

CONDITIONS: Children Who Present to the ED With Minor Febrile Illnesses
Keywords: children; fever; emergency department
MeSH Terms: conditions — Fever; Emergencies | interventions — Methods; Videotape Recording

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): Video (DVD) discharge instructions
  Interventions: Behavioral: Intervention
- Control (No Intervention): Written instructions only

INTERVENTIONS:
Behavioral: Intervention
  Other Names: Video (DVD) discharge instructions
  Arms: Intervention

SUMMARY:
To evaluate the effect of video discharge instructions on return visits to the ER or ED within 72 hours of the original visit for children with febrile illnesses.

DETAILED DESCRIPTION:
This is a randomized prospective convenience study of children presenting to the ED. Children greater than 8 weeks and up to and including their 18th birthday are enrolled. Patients were randomly assigned to one of two study groups: video + written fever specific discharge instructions and only written fever specific discharge instructions. Parents assigned to the video group watched the DVD in the emergency department (ED) and take it home along with the written instructions. At 72 hours both groups received a phone call asking whether they returned to the ED and the usefulness of discharge instructions (DVD and/or written). Critically ill children and those with chronic medical conditions were excluded. The primary outcome is a return ED visit for fever confirmed in our electronic medical record and questionnaire response. The secondary outcome is reported parental usefulness of the discharge instructions.

ELIGIBILITY:
Inclusion Criteria:

* Children ages 8 weeks to 18 years
* Presented to the ED with a chief complaint of fever. Fever was defined as a temperature greater than or equal to 100.4⁰F
* English or Spanish speaking
* Working telephone for follow-up call
* Venue to view DVD at home (TV, computer, etc)

Exclusion Criteria:

* Children with a chronic medical illness
* Children with immune-compromising conditions
* Allergies to acetaminophen or ibuprofen
* Previously enrolled
* Admitted at the time of their index ED visit

Ages: 8 Weeks to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 273 (Actual)
Dates: Start 2011-02 (Actual); Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sharon R Smith, MD, Principal Investigator — Connecticut Children's Medical Center
Locations (1):
- Connecticut Children's Medical Center, Hartford, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Video (DVD) discharge instructions
  Intervention
Period: Overall Study
Arm/Group | Intervention | Control
Started | 140 | 133
Completed | 140 | 133
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 140 | 133 | 273
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 2.7 (3.0) | 2.1 (2.4) | 2.4 (2.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 72 | 74 | 146
  Male | 68 | 59 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 72 | 73 | 145
  Not Hispanic or Latino | 68 | 60 | 128
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 22 | 19 | 41
  White | 31 | 29 | 60
  More than one race | 15 | 13 | 28
  Unknown or Not Reported | 72 | 72 | 144

OUTCOME MEASURES:

1. Primary Outcome: Recidivism
Description: Number of repeat visits to the ED within 72 hours of initial visit for fever
Time Frame: 72 hours
Measure: Number; unit: number of return visits within 72 ho
Arm/Group | Intervention | Control
Number analyzed (Participants) | 140 | 133
number of return visits within 72 ho | 6 | 3

2. Secondary Outcome: Usefulness
Description: Rating of how useful the parents found the discharge instructions
Time Frame: 1 week
Population: Parents were not considered enrolled but contributed to the assessment.
Measure: Number; unit: number of parents found useful
Arm/Group | Intervention | Control
Number analyzed (Participants) | 140 | 133
number of parents found useful | 94 | 94

ADVERSE EVENTS:
Time Frame: Data not collected
Description: All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed.
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes